CLINICAL TRIAL: NCT05790590
Title: Comparison of Image Quality Between "Double Low Dose" Liver CT Using AI-based Iodine Boosting Reconstruction and Standard Contrast-enhanced Liver CT in Patients With Colorectal Cancer: Prospective, Randomized, Non-inferiority Trial
Brief Title: Comparison of Image Quality Between "Double Low Dose" Liver CT and Standard Liver CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: SNUH-2022-3274
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Metastasis to Liver; Colorectal Cancer
Keywords: CT
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dose CT (Active Comparator): Standard dose protocol CT using standard radiation dose (120 kVp) and standard dose of contrast media, and reconstructed with commercially available reconstruction algorithm of the CT scanner.
  Interventions: Diagnostic Test: Standard dose CT
- Double low dose CT (Experimental): Double low dose protocol CT using low radiation dose (120 kVp & 70% of reference mAs of standard dose CT) and low dose of contrast media, and reconstructed with commercially available vendor-agonistic AI-based software.
  Interventions: Diagnostic Test: Double low dose CT

INTERVENTIONS:
Diagnostic Test: Double low dose CT — Simultaneous reduction of both radiation dose and contrast media dose
  Arms: Double low dose CT
Diagnostic Test: Standard dose CT — CT with standard radiation dose and contrast media dose
  Arms: Standard dose CT

SUMMARY:
In patients with malignancies, contrast-enhanced abdominal CT (hereafter abdominal CT) plays an important role in detecting carcinoma recurrence and assessing treatment response. In this study, we aim to investigate whether such a "double low" dose CT is feasible in patients with liver metastases of colorectal cancer using a vendor-agnostic artificial intelligence-based noise reduction and contrast enhancement software.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer (CRC) patients
* on surveillance or monitoring for liver metastasis (of CRC)

Exclusion Criteria:

* any relative or absolute contra-indication of CECT
* diffuse infiltrative type of liver metastasis or on monitoring for too many liver lesions

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
lesion conspicuity on portal venous phase | 6 months after primary study completion.
  qualitative analysis of lesion conspicuity on portal venous phase on five-point scale (higher score indicates better conspicuity).
  Lesion conspicuity is compared between the two arms.

SECONDARY OUTCOMES:
lesion conspicuity on arterial phase | 6 months after primary study completion.
  qualitative analysis of lesion conspicuity on arterial phase on five-point scale (higher score indicates better conspicuity) Lesion conspicuity is compared between the two arms.
lesion detectability | 12 months after primary study completion.
  lesion detectability is compared between the two arms, compared with reference standard. Figure-of-merit was obtained.
Radiation dose | 1 month after primary study completion
  Dose-length product (mGy*cm) is compared between the two arms.
Contrast media (CM) dose | 1 month after primary study completion
  The amount of CM dose is compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No